CLINICAL TRIAL: NCT03067701
Title: Effects of Carbon Monoxide Breathing on Blood Vessel Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro 46208
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2017-10

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carbon Monoxide Inhalation (Experimental): In healthy young adults 18-39 years of age, The Investigator will determine if intermittent inhalation a 0.1% CO, from a 1-liter bag once every minute for 30-40 minutes, at a level that approaches the CO boost with hookah smoking, augments endothelial function, thus implicating CO as the major endothelial vasodilator substance in hookah smoke.
  Interventions: Drug: Carbon Monoxide

INTERVENTIONS:
Drug: Carbon Monoxide — In healthy young adults 18-39 years of age, The investigator will determine if intermittent inhalation of 0.1% CO, from a 1-Liter bag once every minute for 30-40 min at a level that approaches the CO boost with hookah smoking, augments endothelial function.

SUMMARY:
In healthy young adults 18-39 years of age, the investigators will determine if intermittent inhalation a 0.1% CO, from a 1-liter bag once every minute for 30-40 minutes, at a level that approaches the CO boost with hookah smoking, augments endothelial function, thus implicating CO as the major endothelial vasodilator substance in hookah smoke.

Rationale: Our group has demonstrated (PRO36547) that in contrast to cigarette smoking, hookah smoking (tobacco heated with charcoal) acutely augments, rather than impairs, brachial artery FMD. Importantly, our data strongly implicate-but do not prove-that the augmentation in FMD is caused by CO. Therefore; the investigators would like to extend the scientific priority of this work by directly investigating cause and effect of CO breathing (similar levels than ones obtained after hookah smoking) on brachial artery FMD.

DETAILED DESCRIPTION:
Carbon monoxide (CO) is an endogenously produced gas that play important physiological roles in the circulation. Traditionally considered a poisonous gas that causes tissue hypoxia, CO produced by vascular cells as a byproduct of heme catabolism, also functions to regulate blood flow by inhibiting vasomotor tone, smooth muscle cells proliferation, and platelet aggregation. These vascular effects are thought to be mediated by cyclic guanosine monophosphate (cGMP) because both clinical observations and experimental data provide precedent that CO, like nitric oxide, constitutes a cGMP-dependent vasodilator. Drugs that upregulate the endogenous production of CO by heme oxygenase, such as CO releasing molecules (CORMs), are being developed to treat several vascular diseases.

The toxicity of CO is dependent on the dose and duration of exposure. Studies have shown that CO inhalation is fatally toxic at concentrations of 800 parts per million (ppm) or 0.08% in the air. Studies have also demonstrated that CO inhalation at low doses (<250 ppm) offers protection against inflammation and ischemic injury in the heart, liver, and kidney. According to a recent study published in Nature, repeated exposures of 250 ppm of CO for 1 hour inhibit experimental atherosclerosis by a cGMP-dependent process in rats. Other studies have also demonstrated that exogenous CO causes cGMP-dependent vasodilation in isolated vascular rings, and, in intact animals, can augment nitric oxide-dependent vasodilation.

Initial studies by our group allowed us to discover that, in young healthy hookah smokers, hookah smoking is a potent acute stimulus to augment-not impair-endothelial function measured by brachial artery flow mediated dilation (FMD). The data implicate a pivotal mechanistic role of one or more charcoal combustion products in the augmented endothelial function: when burning charcoal was replaced with a healthier electronic heat source ("e-coal"), FMD became acutely impaired just as with cigarettes and almost all other known tobacco products including electronic-cigarettes. Interestingly, the CO boost after our hookah subjects smoked charcoal-heated hookah tobacco was ~10-fold higher than after smoking a cigarette (25+11 vs. 3+2 ppm). Tobacco literature provide evidence that the repeated CO exposure from cigarette smoking is associated with a reduced risk of pre-eclampsia (associated with pathological vasoconstriction) in pregnant women as compared with both non-smokers or users of smokeless tobacco (snuff) which does not generate CO.

Recently published studies by our group showed that sustained CO inhaled by healthy smokers, to achieve mean carboxyhemoglobin 5+1% (which is equivalent to our proposed exhaled CO levels of 35 ppm), had no significant effect on blood pressure, heart rate, plasma catecholamines, platelet aggregation or C-reactive protein, a marker of inflammation. The effects of low levels of CO on human endothelial function has yet to be determined.

Taken all the current evidence together, the present application aims to investigate the acute effects of breathing very low doses CO-to replicate levels obtained with hookah smoking-on peripheral vessel function in humans. the investigators hypothesize that CO is the key charcoal combustion product in hookah smoke that enhances endothelial function, thus masking the impairment seen with hookah tobacco toxicants. The benefit of this amendment is beyond this project, especially if CO inhalation at very low dose, non-toxic levels is shown to decrease cardiovascular risk and augment endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years of age

Exclusion Criteria:

* History of cardiopulmonary, diabetes, dyslipidemia or psychiatric disease
* BP > 140/90 mmHg
* BMI <18.5 or > 30 kg·m2
* Resting heart rate > 100 beats/min
* Taking prescription medication
* Hemoglobin levels < 11.6 g/dL
* Total cholesterol > 240 or HDL < 36
* Fasting glucose >100 mg/dL or <60 mg/dL
* Bilirubin >1.2 mg/dL; albumin < 3.5 or > 5.5 g/dL; alkaline phosphatase (alk phos) >125 IU/L; alanine aminotransferase (ALT) > 45 U/L; aspartate aminotransferase (AST) > 35 U/L
* Positive (+) toxicology screen
* Pregnant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
To determine the effect of intermittent inhalation of 0.1% CO from 1-liter bags on endothelial function measured by brachial artery flow mediated dilation. | immediate assessment of endothelial function measured by brachial artery flow-mediated dilation after 30-40 minutes of adminstration
  assessment of endothelial function measured by brachial artery flow-mediated dilation after 30-40 minutes of carbon monoxide adminstration

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Director, Hypertension Center Associate Director, Cedars-Sinai Heart Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezk-Hanna M, Mosenifar Z, Benowitz NL, Rader F, Rashid M, Davoren K, Moy NB, Doering L, Robbins W, Sarna L, Li N, Chang LC, Elashoff RM, Victor RG. High Carbon Monoxide Levels from Charcoal Combustion Mask Acute Endothelial Dysfunction Induced by Hookah (Waterpipe) Smoking in Young Adults. Circulation. 2019 May 7;139(19):2215-2224. doi: 10.1161/CIRCULATIONAHA.118.037375. PMID 30764644